CLINICAL TRIAL: NCT05807815
Title: Determination of the Incidence of Hyperoxia and the Effectiveness of FiO2 Titration Guided by the Oxygen Reserve Index in Preventing Hyperoxia in Mechanically Ventilated Patients in the Intensive Care Unit.
Brief Title: The Effectiveness of the Use of Oxygen Reserve Index in Preventing Hyperoxia in the Intensive Care Unit.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aykut Saritas, associated professor, Tepecik Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Health Sciences University
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Hyperoxia; Complication; Mechanical Ventilation Complication
Keywords: Hyperoxia; Fraction of inspired oxygen; Intensive care unit
MeSH Terms: conditions — Hyperoxia | interventions — Oxygen Saturation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Patients with oxygen saturation > 97% will only be observed. ORi values will be recorded blindly from the clinician. Adjustments to be made in FiO2 will be determined by the intensive care doctor independently of the study, and only observation will be made in this group.
- ORi+SpO2 (oxygen saturation) group (Active Comparator): Fraction of inspired oxygen (FiO2) is titrated guided by oxygen saturation in that range; %95<oxygen saturation≤%98
  Interventions: Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and oxygen saturation

INTERVENTIONS:
Procedure: Titration of fraction of inspired oxygen (FiO2) guided by ORI and oxygen saturation — FiO2 will be titrated by reducing 10% if Ori>0.01 and oxygen saturation ≥ 98% until Ori is 0.00.
  FiO2 will not be changed if Ori is 0.00 and %95<oxygen saturation≤%98 FiO2 will be increased by 10% if oxygen saturation <95 or PaO2<60 mmHg
  Arms: ORi+SpO2 (oxygen saturation) group

SUMMARY:
Oxygen therapy is the most common treatment modality for patients with hypoxemia in intensive care units, but target values for normoxemia are not clearly defined. Therefore, iatrogenic hyperoxemia is a very common situation. In intensive care units, FiO2 is usually adjusted according to hypoxia and hyperoxia is ignored in patients under mechanical ventilator support. Even though there are many side effects reported related to hyperoxemia and hyperoxemia is shown to be related to worse outcome than expected; clinicians still observe hyperoxemia frequently.

Continuous ORi monitoring can be used for detecting and preventing hyperoxia. The ability to perform FiO2 titration with ORi may be an appropriate monitoring management to prevent the harmful effects of hyperoxia. In this study, it was aimed to investigate the effectiveness of ORi-guided FiO2 titration in preventing hyperoxia in patients undergoing mechanical ventilation in the intensive care unit and to determine the incidence of hyperoxia.

DETAILED DESCRIPTION:
In intensive care units, FiO2 is usually adjusted according to hypoxia and hyperoxia is ignored in patients under mechanical ventilator support. Even though there are many side effects reported related to hyperoxemia and hyperoxemia is shown to be related to worse outcome than expected; clinicians still observe hyperoxemia frequently.

Oxygen reserve index (ORi™) (Masimo Corp., Irvine, USA) can guide clinicians in detection of hyperoxia. ORi is a parameter which can evaluate partial pressure of oxygen (PaO2) rating from 0 to 1. There are growing evidences in ORi that it might be helpful to reduce hyperoxia in general anesthesia. Continuous ORi monitoring can be used for detecting and preventing hyperoxia. The ability to perform FiO2 titration with ORi may be an appropriate monitoring management to prevent the harmful effects of hyperoxia.

In this study, it was aimed to investigate the effectiveness of ORi-guided FiO2 titration in preventing hyperoxia in patients undergoing mechanical ventilation in the intensive care unit and to determine the incidence of hyperoxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years,
* Patients whose oxygen saturation >97%
* Patients that have invasive arterial monitorization

Exclusion Criteria:

* Patients younger than 18
* Patients that need to be treated with high doses of vasopressors,
* Patients having peripheric hypoperfusion,
* Hemodynamically unstable patients,
* Patients with hemoglobinopathy,
* Pregnancy,
* Morbid obesity (bmi>40 kg/m2),
* Patients with arrythmia that can result in hemodynamic instability, patients with acute coronary syndrome
* Acute respiratory failure or ARDS.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Correlation of FiO2 and ORi value | Up to 24 weeks
  Correlation of FiO2 value and ORi value. FiO2 adjusted until ORi reaches to zero and %95<oxygen saturation≤%98

SECONDARY OUTCOMES:
Fraction of inspired oxygen (FiO2) | Up to 48 hours
  Fraction of inspired oxygen (FiO2) in every 4 hour intervals
Mean arterial blood pressure (MAP) | Up to 48 hours
  Measurement of mean arteria blood pressure (SBP)
Heart rate (HR) | Up to 48 hours
  Measurement of heart rate (HR)
Positive end-expiratory pressure (PEEP) | Up to 48 hours
  Measurement of PEEP

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Konak, Turkey (Türkiye)

REFERENCES:
- [Background] de Graaff AE, Dongelmans DA, Binnekade JM, de Jonge E. Clinicians' response to hyperoxia in ventilated patients in a Dutch ICU depends on the level of FiO2. Intensive Care Med. 2011 Jan;37(1):46-51. doi: 10.1007/s00134-010-2025-z. Epub 2010 Sep 28. PMID 20878146
- [Background] Rincon F, Kang J, Maltenfort M, Vibbert M, Urtecho J, Athar MK, Jallo J, Pineda CC, Tzeng D, McBride W, Bell R. Association between hyperoxia and mortality after stroke: a multicenter cohort study. Crit Care Med. 2014 Feb;42(2):387-96. doi: 10.1097/CCM.0b013e3182a27732. PMID 24164953
- [Background] Mach WJ, Thimmesch AR, Pierce JT, Pierce JD. Consequences of hyperoxia and the toxicity of oxygen in the lung. Nurs Res Pract. 2011;2011:260482. doi: 10.1155/2011/260482. Epub 2011 Jun 5. PMID 21994818
- [Background] Scheeren TWL, Belda FJ, Perel A. Correction to: The oxygen reserve index (ORI): a new tool to monitor oxygen therapy. J Clin Monit Comput. 2018 Jun;32(3):579-580. doi: 10.1007/s10877-018-0104-9. PMID 29445905
- [Background] Yoshida K, Isosu T, Noji Y, Ebana H, Honda J, Sanbe N, Obara S, Murakawa M. Adjustment of oxygen reserve index (ORi) to avoid excessive hyperoxia during general anesthesia. J Clin Monit Comput. 2020 Jun;34(3):509-514. doi: 10.1007/s10877-019-00341-9. Epub 2019 Jun 22. PMID 31227971